CLINICAL TRIAL: NCT07224256
Title: VOICE: An Early Feasibility Study of a Precise Robotically Implanted Brain-Computer Interface for Communication Restoration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuralink Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: N1-EFS-200
Record Dates: First submitted 2025-10-13; First posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Tetraplegia/Tetraparesis; Quadriplegia; Cervical Spinal Cord Injury; Amyotrophic Lateral Sclerosis; Quadriplegia/Tetraplegia; Tetraplegic; Paralysis; Stroke
Keywords: stroke; spinal cord injury; SCI; ALS; brain computer interface; BCI; PLS; voice; speech; dysarthria; neuralink
MeSH Terms: conditions — Quadriplegia; Amyotrophic Lateral Sclerosis; Paralysis; Stroke; Spinal Cord Injuries; Speech; Dysarthria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Neuralink N1 Implant and R1 Robot (Experimental): Implantation of the N1 Implant by the R1 Robot.
  Interventions: Device: N1 Implant; Device: R1 Robot

INTERVENTIONS:
Device: N1 Implant — The N1 Implant is a type of implantable brain-computer interface
  Other Names: Neuralink N1 Implant, N1, Telepathy, Link
Device: R1 Robot — The R1 Robot is a robotic electrode thread inserter that implants the N1 Implant.
  Other Names: R1, Neuralink R1 Robot

SUMMARY:
The VOICE Study is an early feasibility study to evaluate the initial clinical safety and efficacy of the N1 and R1 Systems device design concept in providing an ability to communicate. The Neuralink N1 Implant is intended to provide the ability to communicate to individuals with severe and irreversible speech production impairment. It is indicated for adults with neurological conditions of the central speech pathways who have impaired upper limb function. The N1 Implant is a skull-mounted, wireless, rechargeable implant connected to electrode threads that are implanted in the brain by the R1 Robot, a robotic electrode thread inserter.

ELIGIBILITY:
Inclusion Criteria:

Adults with diagnosis of ALS, PLS, stroke, or Spinal Cord Injury who have severe speech impairment and impaired upper limb function.

* Life expectancy ≥ 12 months.
* Ability to communicate in English
* Presence of a stable caregiver

Exclusion Criteria

* Moderate to high risk for serious perioperative adverse events
* Morbid obesity (Body Mass Index > 40)
* History of poorly controlled seizures or epilepsy
* History of poorly controlled diabetes
* Requires magnetic resonance imaging (MRI) for any ongoing medical conditions
* Acquired or hereditary immunosuppression
* Psychiatric or psychological disorder
* Brain MRI demonstrating hemorrhage, tumor, distorted or adverse anatomy.
* Any condition which, in the opinion of the Investigator, would compromise your ability to safely participate in the study or undergo the implantation procedure

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Device-Related Adverse Events (AE) | 12 months post-implant
  The proportion of subjects with device-related adverse events (AEs) at the 12-month follow-up visit.
Procedure-Related Adverse Events (AE) | 12 months post-implant
  The proportion of subjects with procedure-related adverse events (AEs) at the 12-month follow-up visit.

SECONDARY OUTCOMES:
Long-term Device-Related Adverse Events (AE) | Up to 48 months post-implant
  The proportion of subjects with device-related adverse events (AEs) up to the 48-month long-term follow-up visit.
Long-term Procedure-Related Adverse Events (AE) | Up to 48 months post-implant
  The proportion of subjects with procedure-related adverse events (AEs) up to the 48-month follow-up visit.
Preliminary efficacy of the R1 Robot | During surgical implantation procedure
  Preliminary efficacy of the R1 Robot will be evaluated by measuring the following percent of electrodes inserted (reported as electrodes inserted / total electrodes).
Preliminary efficacy of the N1 Implant | Up to 48 months post-implant
  Preliminary efficacy of the N1 Implant will be evaluated by measuring the following BCI performance for speech, quantified by measuring the monthly maximum correct word per minute (CWPM).

CONTACTS AND LOCATIONS:
Overall Officials: Nader Pouratian, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: https://neuralink.com/ — https://neuralink.com/